CLINICAL TRIAL: NCT06073392
Title: The Effect of the Different Number of Topics in Educational Video on Oral Health Status of Preschool Children: Study Protocol for a Cluster Randomized Controlled Trial (RCT)
Brief Title: Cluster RCT on the Effect of the Topics Number in Oral Health Educational Video Among Preschool Children.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, SITI NUR BAIDURI BINTI MOHD JAINI, Principle Investigator, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: USM/JEPeM/KK/23060506; NMRR ID-23-01742-04F (Registry Identifier: National Medical Research Registration)
Record Dates: First submitted 2023-10-03; First posted 2023-10-10 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Oral Health
Keywords: oral health; oral hygiene; dental plaque; gingivitis; child
MeSH Terms: conditions — Dental Plaque; Gingivitis

STUDY DESIGN:
Intervention Model Description: Model is multiple-arm parallel group. There are multiple-arm trials, four experimental are versus single-control arm.
  Four experimental arms intervention are:
  1. effective toothbrushing technique (1 topic)
  2. effective toothbrushing technique, effects of sugary diet (2 topics)
  3. effective toothbrushing technique, and dental caries (2 topics)
  4. effective toothbrushing technique, effects of sugary diet, and dental caries (3 topics)
  Single placebo arms is topic on tooth anatomy and eruption
Who Masked: Participant
Masking Description: Masking: Single-blinded, where participants are unaware of the type of intervention given to them (in which combination and either 1 topics, 2 topics or 3 topics)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intervention Group 1 (IG1) (Experimental): Subjects in IG1 will be given a animation video screening in a specific room. IG1 intervention is on one topic cover only. The animation educational video covers on the topic of effective toothbrushing technique.
  Interventions: Other: Educational video
- Intervention Group 2 (IG2) (Experimental): Subjects in IG2 will be given a animation video screening in a specific room. IG2 intervention is on two topics cover only. The animation educational video covers on the topic of effective toothbrushing technique and effects of sugary diet.
  Interventions: Other: Educational video
- Intervention Group 3 (IG3) (Experimental): Subjects in IG3 will be given a animation video screening in a specific room. IG3 intervention is on two topics cover only. The animation educational video covers on the topic of effective toothbrushing technique, and dental caries.
  Interventions: Other: Educational video
- Intervention Group 4 (IG4) (Experimental): Subjects in IG4 will be given a animation video screening in a specific room. IG4 intervention is on three topics cover. The animation educational video covers on the topic of effective toothbrushing technique, effects of sugary diet, and dental caries.
  Interventions: Other: Educational video

INTERVENTIONS:
Other: Educational video — Educational video in animation mode

SUMMARY:
Purpose: This cluster randomized controlled trials study aims to investigate whether different number of topics delivered through educational video affect the oral health status, knowledge, attitude and practice of preschool children.

Hypothesis: The hypothesis of this study is the number of topics covered in educational videos aimed at preschool children will have a direct impact on their oral health status.

The specific hypothesis is the educational videos covering wide range of oral health topics will lead to better oral health outcomes in preschool children compared to videos focusing on limited number of topics. The higher number of topics delivered in educational video, the better oral health status, knowledge, attitude, and practice.

The alternative hypothesis is the combination of three topics on effective toothbrushing technique, effects of sugary food, and dental caries is effective to led to the most improvement in oral health status, knowledge, attitudes, and practices compared to two or only one topic.

Objectives: The objectives of this study were divided into primary and secondary.

The primary objective of the study is to assess the effect of different number of topics in educational video versus placebo video on mean difference in plaque score and gingival score among preschool children at baseline and 4 weeks after intervention.

The secondary objective is to assess the effect of different number of topics in educational video versus placebo video on mean difference in knowledge, attitude and practice score among preschool children at baseline and 4 weeks after intervention.

Participants: The study will involve 124 preschool children aged five to six years old.

Methods: Researchers will randomize classes in the school into five clusters using closed enveloped technique. These five clusters will be randomly assigned either into interventional groups or control groups. There are four intervention groups and one control group. Each intervention group will be compared to a control group for mean difference in plaque, gingival and KAP score at baseline and after intervention.

Duration: The study is expected to last 6 months (from subjects recruitment to final research report) with regular updates on progress.

Location: The study will be conducted at a preschool in Kota Bharu Kelantan.

DETAILED DESCRIPTION:
Study Design:

This is the phase I interventional cluster randomized controlled trial with multiple-arm parallel group assignment and single blinded masking for prevention of dental caries and gingivitis among preschool children.

The rationale of using this design because it is suitable for preschool-level and logistically simpler. Besides that, this design can minimize the risk of contamination and also resemble the real-word applicability of the program.

Study population:

Preschool children in Kota Bharu, Kelantan

Participants:

The participants are preschool children aged 5 to 6 years old. One preschool will be involved in this study. The reason behind the selection of this school is because of the availability of multiple classes at one. There are about 240 students distributed across 10 classes or 24 students per class on average. There are five classes for five years old and five classes for six years old children. All students will be invited to participate in the study.

Out of five groups, four groups are for intervention and one group is for control. Participants will be asked to watch educational videos about oral health as the intervention material in this study. The participants will be divided into five groups according to type of intervention whether to watch video with one, two or three topics as below:

* Group 1: toothbrushing technique topic only (1 topic)
* Group 2: combination of toothbrushing technique and sugary diet (2 topics)
* Group 3: combination of toothbrushing technique and dental caries (2 topics)
* Group 4: combination of toothbrushing technique, sugary diet and dental caries (3 topics)
* Group 5: no intervention (no video show will be provided)

Researchers will compare oral health, knowledge, attitude and practice score at baseline and after intervention within each group. Researchers also will compare the mean difference of oral health, knowledge, attitude and practice score between intervention group and control group.

Randomization:

A cluster randomization sampling method will be used because of the age-segregated school system. Then, the classes from each age strata will be randomly allocated into five groups using sealed enveloped technique. At the end, each group consists of two classes, one from the five-year-old class and another one from six years old class. The sample in each group will be equally distributed between five years old and six-year-old class. Based on calculated sample size, 25 students needed for each group. 12 students of five years old and 13 students of six years old will be randomly selected as subjects in each group.

Interventions:

The educational videos that will be used as intervention are in animation design, with a duration of maximum six minutes for each video. Videos used are from the existing resources that used my Ministry of Health, Malaysia (oral health program) to preschool children. Topics that will be covered are effective toothbrushing techniques, the effects of sugary diet and literacy on dental caries. Each of the topics will be covered in a separate video. The video will be merged according to the intervention group requirement in intervention process.

Data collection:

The procedure involving questionnaire distribution and video show will be conducted in the specific identified room. Health room (Bilik Kesihatan) has been identified as the location to conduct the guided questionnaire session and video show session. The guided questionnaire session will be conducted in a small group (25 students each session). As for the video screening, it will be conducted to involve all students in the class involved.

The intervention will be conducted in the Bilik Kesihatan. Students in classes under control group will not be given any educational video screening during study period.

Ethical Considerations:

All study procedure to be carried out in a non-invasive manner and will be using non-invasive instruments. The approval of the ethics committee, main supervisor and co-supervisors is obtained before the questionnaire is distributed to all respondents. Subjects will not be named in subsequent write-ups and materials submitted for publication. Ethical approval to conduct this study will be obtained from the Human Research Ethics Committee of Universiti Sains Malaysia and National Medical Research Register, Ministry of Health Malaysia.

The general procedures for obtaining informed consent from parents and preschool children is begin with the initial contact by contacting the preschool and explain the purpose and nature of the study, as well as its potential impact on the preschool and its students. Following that, the written proposal prepared to outline the plan to involve the preschool in the research. Then, meetings will be conducted with preschool administrators, teachers, and staff to discuss the study further and to distribute the informed consent form to the parents of preschool children through class teacher. A letter to parents of preschool-aged children attached together with the patient Information Sheet (PIS) and the informed consent form. The child's participation is voluntary, and parents' consent is required.

Data Analysis:

Data collected in the study will be entered and analyzed using IBM SPSS. Descriptive analysis will be used for the socio-demographic characteristics, including the children's age, sex, race, caregivers' education level and household income in the control and intervention groups. Paired t-test will be used for the comparison within groups in the mean dental plaque score and in mean KAP score before and after the intervention. Analysis of covariance (ANCOVA) will be used for the comparison between groups in the difference in dental plaque score adjusted for difference in KAP score.

Timeline:

i. Recruitment of subject: 2 weeks ii. Baseline data collection

* Questionnaire: 1 week
* Oral screening: 1 week iii. Intervention (video show screening): 1 week iv. Post intervention waiting period data collection post intervention period : 4 weeks v. Post intervention data collection
* Questionnaire : 1 week
* Oral screening: 1 week vi. TOTAL = 11 weeks

Sample Size and Power Analysis:

The effect size included is 0.51 to inflate the individual randomization in this stratified cluster study design. The total number of samples is n=103 with 21 subjects per group). The total sample size after accounting for 20% dropouts is 124 or 25 subjects per group.

Potential Challenges:

Cluster-level variation may arise among preschools children in terms of infrastructure, resources, and practices which can impact the effectiveness of the interventions. It can be minimized by selecting one school consisting of a larger number of classes and students under management.

The risk of contamination between intervention and control groups within the same preschool can occur if children interact with each other, potentially diluting the treatment effect. Therefore, intervention will be given in groups within each class member in order to minimize the contamination between groups of interventions as well as control group.

Preschool children may not consistently attend the school, leading to missing data and potential attrition bias. Data collection may be extended to cather all subjects. Honorarium provided to motivate participation throughout the study period.

ELIGIBILITY:
Inclusion Criteria:

* Children aged five to six years old and understand the Malay language.
* Children with normal cognitive and psychomotor ability equal to normal children aged five to six years old
* Children who unable to read and write fluently but able to understand instructions

Exclusion Criteria:

* Children with physical and psychological condition that prevents them from understanding and following the instruction.

Ages: 5 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 125 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Plaque score using Modified Dental Plaque (MPI) | Baseline and 4 weeks after intervention
  The index will be calculate dental plaque on each tooth surface. The MPI score is obtained by the sum of the plaque score for all teeth, divided by the number of surfaces scored.
  Minimum value for the score is 0, while the maximum value is 5. The higher the score value describes the more plaque accumulation on each subject. Therefore, a high plaque score is interpreted as poor oral hygiene status.
  To give clinical relevance to the index, the index translated into four oral hygiene categories as 0 - 1.25: Excellent, 1.25 - 2.50: Good, 2.50 - 3.75: Fair, 3.75 - 5.00: Poor
Gingival Score using Modified Gingivitis Plaque (MGI) | Baseline and 4 weeks after intervention
  The index will be calculated the extent and the severity of gingival inflammation using four ordinals.
  The MGI score is obtained by the sum of the gingival score for all teeth, divided by the number of surfaces scored.
  The minimum value for the score is 0, while the maximum value is 3. The higher the score value describes the more severe inflammation due to plaque accumulation in subject. Therefore, a high gingival score is interpreted as poor gingival health. To give clinical relevance to the index, the index translated into three gingivitis categories, 0 : No gingivitis, ≤1.0 : Mild gingivitis, ≤2.0 : Moderate gingivitis, ≤3.0 : Severe gingivitis.

SECONDARY OUTCOMES:
Knowledge, Attitude, Practice (KAP) level using KAP score | Baseline and 4 weeks after intervention
  KAP score generated from the validated questionnaire used in National Oral Health Survey of Preschool Children, Ministry of Health, Malaysia, 2015. Response options are binary in nature, as the question for preschool children is age-appropriate language that preschool children can comprehend with a straightforward and factual answer. This questionnaire will be validated for content and response process. The questionnaire consists of three domains with 18 items. The domains are knowledge (6 items), attitude (6 items) and practice (6 items). Total score of knowledge, attitude and practice (6X3) is 18. Each item will be given with responses 'Yes' and 'No'. Each item is assessed by one correct answer from answer options with total KAP score ranged from 0 to 18. Average score will be translated into percentage. Then, the score translated into three KAP level categories as, <30%: Poor OHKAP, 30% - 60%: Fair OHKAP, > 60% Good OHKAP

CONTACTS AND LOCATIONS:
Overall Officials: SITI NUR BAIDURI MOHD JAINI, Principal Investigator — SCHOOL OF DENTAL SCIENCES, UNIVERSITI SAINS MALAYSIA

IPD SHARING:
Plan to Share IPD: No
Data will be shared with qualified researchers upon request, subject to ethical and legal considerations, and after the approval of a data sharing agreement. Data sharing is subject to restrictions that include a 12-month embargo period following publication and a prohibition on using the data for commercial purposes. Before sharing, all individual participant data will be de-identified to protect privacy. Any potentially identifying information will be removed or altered. Data sharing will be conducted in accordance with the ethical guidelines set forth by Human Research Ethics Committee USM and in compliance with relevant data protection laws, including Personal Data Protection Act 2010